CLINICAL TRIAL: NCT04490291
Title: An Observational Study of Integrated Chronic Pain Management in a Community Health Center
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Logan University (Unknown)
Responsible Party: Principal Investigator, Chrisotpher Prater, Assistant Professor in Medicine and Pediatrics, Washington University School of Medicine
Other Study IDs: RD04240531
Record Dates: First submitted 2020-06-17; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain; Spine Disease
Keywords: community health center; integrated pain team
MeSH Terms: conditions — Chronic Pain; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: chronic pain team — enrollment in chronic pain team at study site
Other: chiropractic team — enrollment in chiropractic team/intervention at study site

SUMMARY:
This was a prospective observational study with the primary objective of quantifying a change in pain scores after 6-12 months of two separate interventions within the study site (pain team and chiropractic team). Target enrollment was 30 participants for each intervention. The primary outcome was a change from baseline of the Pain Disability Questionnaire (PDQ), the study tool. Secondary outcomes were reduction of opioid dose by morphine equivalent daily dose, and its effect on PDQ scores.

DETAILED DESCRIPTION:
Data collection After participants were enrolled, they completed a baseline PDQ while waiting for their appointment. Participants continued to see the intervention group, PCP, and other medical providers as determined by their health providers independent of this study's protocol. Another PDQ was collected at an intended 6 - 12 months later. Demographic information was collected by manual chart review in the electronic medical record NextGen (NextGen EHR, Nextgen Healthcare, Inc. Irvine, CA, USA).

Variables collected included age, sex, race, BMI, insurance type, preferred language, presence of another pain diagnosis (e.g. knee pain), active mental health diagnosis (including substance abuse), diagnosis of hypertension or diabetes, and morphine equivalent dose (MED); one post-hoc variable was recorded: timing of follow-up survey in relation to the 2019 coronavirus (COVID-19) pandemic, defined as before/after March 1, 2020. Intervention type was analyzed as an independent variable since the study was not designed as a comparison of interventions. All data was stored in an encrypted Excel database on a password-protected laptop. Consent forms were stored in a locked cabinet accessible only to the PI.

Stata 16.0 (StataCorp, LLC, College Station, TX, USA) was used for statistical analysis. PDQ scores at baseline and follow-up were tested for statistical significance using paired t-tests. Univariate analysis was performed on individual categorical variables and change in PDQ using two-sample t-tests. Multivariate linear regression was used to determine associations of these factors to the outcome. Variables were excluded from regression models if there was a subgroup size of six or less.

ELIGIBILITY:
Inclusion Criteria:

* referred by PCP to either intervention at study site

Exclusion Criteria:

* active cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: active patients at an urban federally-qualified health center
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
change in Pain Disability Questionnaire (PDQ) score | 6-12 month
  6-12 month follow up pain score - (minus) baseline. scores range from 0 (no pain or disability) to 150 (severe pain and disability)

SECONDARY OUTCOMES:
prescription opioid weaning | 6-12 months
  ability to successfully wean off opioid prescription

CONTACTS AND LOCATIONS:
Locations (1):
- Affinia Healthcare, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
methodology and data will be available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after publication, available indefinitely
Access Criteria: by request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04490291/Prot_SAP_000.pdf